CLINICAL TRIAL: NCT01364935
Title: Pilot Study Comparing Fertility Monitors: DuoFertility Monitor, LadyComp/Babycomp Monitor and Clearblue Ovulation Tests in Support of FDA Application
Brief Title: Comparison of DuoFertility, LadyComp/BabyComp and Clearblue Monitors
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Cambridge Temperature Concepts (Industry)
Responsible Party: Principal Investigator, Joanne Outtrim, RN, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A092165; 11/EE/0016 (Other: National Research Ethics Committee); NCT01343199 (obsolete NCT alias)
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparative study to determine whether several fertility monitoring products - the DuoFertility monitor, the LadyComp/Babycomp monitor and Clearblue Ovulation tests - are substantially equivalent in performance, and secondarily to determine the appropriateness of labeling information for the DuoFertility monitor.

DETAILED DESCRIPTION:
The investigators plan to recruit 30 women who are currently trying to conceive, and ask them to use the 3 fertility monitors for duration of 3 menstrual cycles. Additionally, during the study the women will be asked to fill in online questionnaires to assess the usability of the monitors. As the spouse is often a critical partner in the purchase decision and compliance, the investigators will also ask the spouse to complete similar online questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation
* Females aged 18 to 44 years
* Have a body mass index (BMI) above 19 and below 29
* Regular menstrual cycles, i.e. no greater than 7 days difference between the shortest and longest cycle in the last 6 months
* Minimum menstrual cycle 24 days
* Maximum menstrual cycle 33 days
* Female participants willing to use the 3 fertility monitors for at least 3 cycles.
* Willing to fill in regular questionnaires and study diaries

Exclusion Criteria:

* Women aged younger than 18 years, or older than 44 years
* Have a BMI less than 18 or greater than 29
* Any diagnosed systemic illnesses, including but not restricted to thyroid disease, diabetes or inflammatory diseases
* Polycystic ovary disease
* Endometriosis or other pelvic pathology (including proven tubal disease)
* Taking steroids, including oral contraceptives or anti inflammatory drugs

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female participants trying to conceive, with regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basil Matta, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom